CLINICAL TRIAL: NCT01660243
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Fixed-dose, Parallel-group, Multicenter, Efficacy, and Safety Study of MT-9938 for Treatment of Uremic Pruritus in Subjects With End-stage Renal Disease Receiving Hemodialysis
Brief Title: Efficacy and Safety of MT-9938 for Treatment of Uremic Pruritus in Subjects With End-stage Renal Disease Receiving Hemodialysis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study has been terminated because of insufficient patient recruitment.
Sponsor: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT-9938-A01
Record Dates: First submitted 2012-08-02; First posted 2012-08-08 (Estimated); Results first posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2021-11

CONDITIONS: Uremic Pruritus
Keywords: Pruritus; Renal dialysis; Receptors, Opioid, kappa; Sleep Disorders; Quality of Life
MeSH Terms: conditions — Pruritus; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MT-9938 2.5μg (Active Comparator)
  Interventions: Drug: Nalfurafine hydrochloride(MT-9938) 2.5μg
- MT-9938 5μg (Active Comparator)
  Interventions: Drug: Nalfurafine hydrochloride(MT-9938) 5μg
- MT-9938 10μg (Active Comparator)
  Interventions: Drug: Nalfurafine hydrochloride(MT-9938) 10μg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nalfurafine hydrochloride(MT-9938) 2.5μg — 2.5 μg (2capsules) once daily for 8 weeks
  Arms: MT-9938 2.5μg
Drug: Nalfurafine hydrochloride(MT-9938) 5μg — 5 μg (2capsules) once daily for 8 weeks
  Arms: MT-9938 5μg
Drug: Nalfurafine hydrochloride(MT-9938) 10μg — 10 μg (2capsules) once daily for 8 weeks
  Arms: MT-9938 10μg
Drug: Placebo — Placebo (2capsules) once daily for 8 weeks
  Arms: Placebo

SUMMARY:
This study is being conducted to investigate the efficacy of MT-9938 compared with placebo after 2 weeks, to continue to evaluate efficacy for an additional 6 weeks, and to explore the effect of a reduction in itching intensity on health-related Quality of Life(QoL) domains, especially those which recent research suggests have a positive correlation with overall survival for this patient group. The study will consist of the following phases: Screening (1 to 2 weeks), Run in (1 week), double-blind Treatment (8 weeks), Washout (1 week) culminating in a Follow-up Visit (1 week after the last dose).

DETAILED DESCRIPTION:
This study has been terminated because of insufficient patient recruitment. There were no safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* On stable hemodialysis for at least 3 months
* Has stable functioning arteriovenous fistula, graft or other venous access
* Has continued (uncontrolled) uremic pruritus despite standard of care in the institution
* Has severe pruritus, as determined by a qualifying score of ≥3 on the Itch Severity Score Scale (0 to 4) either day or night during the week prior to Screening Visit
* Has no known drug addiction to any prescription, nonprescription, herbal or natural drugs, and successfully passes a drug screen test
* Women and men whose partners are of childbearing potential agree to practice the medically acceptable methods of birth control and agree to continue with the regimen throughout the duration of the study
* Capable of understanding and responding to the subject questionnaires, understands the purpose and risks of the study, and has given written informed consent
* Has rated his/her NRS score each day for at least 5 days out of the 7 days of the Run-in Phase
* Has severe pruritus, as determined by qualifying mean worst NRS score in a day of ≥5 (on 11 point NRS) at the end of the 1-week Run-in Phase

Exclusion Criteria:

* Current, clinically significant medical comorbidities
* Abnormal liver dysfunction
* Pruritus attributed mainly to any disease unrelated to kidney disease
* Calcium x phosphorus product >80 mg2/dL2 or hemoglobin <7 g/dL or parathyroid hormone levels >1000 pg/mL at Screening
* Received ultraviolet B treatment within 30 days prior to Screening
* Started or changed psychotropic medication within 14 days prior to Screening
* Is receiving opioid antagonists or opioid agonists within 7 days prior to Screening and not willing to abstain from these medications during the study.
* Started or changed medications, creams or emollients including over-the-counter oil bath treatment for relief of pruritus within 7 days prior to Screening
* Has known hypersensitivity to opioids or the study drug ingredients
* Is currently participating in an investigational drug or device clinical study or was participating in such a study within 30 days prior to the start of Screening
* Female subject who is known to be pregnant or nursing
* Is considered not suitable for inclusion in the study in the opinion of Investigator
* Has current suicidal ideation with some intent to act or with specific plan and intent or had suicidal behavior at any time in subject's life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Los Angeles, California
  - New York, New York
  - Rosedale, New York
  - San Antonio, Texas

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who remained eligible entered the 1-week Run-in Phase. The NRS, VAS, and Itch Severity Score were averaged and formed the Baseline itch-intensity scores.
  After the Run-in, subjects who met additional inclusion criteria (having an NRS score for at least 5 days out of the 7 days and a mean worst NRS score ≥5) entered the Double-blind Treatment Phase (8 weeks) and were randomized to 1 of 4 study treatments.
Period: Overall Study
Arm/Group | MT-9938 2.5μg | MT-9938 5μg | MT-9938 10μg | Placebo
Started | 10 | 13 | 11 | 11
Completed | 8 | 13 | 9 | 10
Not Completed | 2 | 0 | 2 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Unable to visit clinic to obtain study drug due to hospitalization | 1 | 0 | 0 | 0
Not completed — Subject was noncompliant with study drug after experiencing AEs; was not discontinued due to the AEs | 0 | 0 | 1 | 0
Not completed — Randomization error | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | MT-9938 2.5μg | MT-9938 5μg | MT-9938 10μg | Placebo | Total
Number analyzed (Participants) | 10 | 13 | 11 | 11 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (10.62) | 54.6 (12.78) | 55.3 (13.64) | 55.2 (12.94) | 55.8 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 4 | 13
  Male | 5 | 11 | 9 | 7 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Worst-itching 11-point Numerical Rating Scale (NRS)
Description: The subject indicated the number on the line from left (0:no itching) to right (10:worst itch I have ever experienced). Assessments was made twice daily using an electronic Patient Reported Outcomes (ePRO) device from the Screening Visit to the Follow-up Visit (Week 9). The 2 daily assessments was separated by 12 h, at approximately 8 am and at approximately 8 pm. Subjects selected the number that best described the worst itch during the day (assessed at approximately 8 pm) or during the night (assessed at approximately 8 am). The day or night score, whichever was greater, was used to calculate the weekly average score and changes from baseline (average over the Run-in Phase [Days -7 to -1]) score in weekly average at 2, 4 and 8 weeks as specified in the protocol are reported. Amount of change score of plus indicates worsening, and minus indicates improvement.
Time Frame: 2 weeks, 4 weeks and 8 week
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MT-9938 2.5μg | MT-9938 5μg | MT-9938 10μg | Placebo
Number analyzed (Participants) | 10 | 13 | 11 | 11
score on a scale
  At 2 weeks | -1.11 (1.224) | -1.19 (1.177) | -1.12 (0.828) | -2.27 (2.774)
  At 4 weeks | -1.41 (2.032) | -2.12 (2.527) | -1.85 (1.392) | -2.25 (3.114)
  At 8 weeks (EOT) | -2.33 (2.269) | -3.13 (2.833) | -3.42 (2.262) | -3.39 (3.614)

2. Primary Outcome: Change From Baseline in Worst-itching Visual Analog Scale (VAS)
Description: The subject placed a single vertical mark on the line of a VAS corresponding to degree of itching intensity from left (no itching) to right (worst itch I have ever experienced). The VAS represents a 100 mm line. It consists of 101 selectable regions and the subject's score on the VAS will correspond to the region (0 to 100) selected on the line. Assessments was made twice daily using an ePRO device from the Screening Visit to the Follow-up Visit (Week 9). The 2 daily assessments was separated by 12 h, in the morning at approximately 8 am and in the night at approximately 8 pm. Subjects put a single vertical mark on the line to show the intensity of your worst itching during the day or during the night. The day or night score, whichever was greater, was used to calculate the weekly average score and changes from baseline in weekly average at 2, 4 and 8 weeks as specified in the protocol are reported. Amount of change score of plus indicates worsening, and minus indicates improvement.
Time Frame: 2 weeks, 4 weeks and 8 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MT-9938 2.5μg | MT-9938 5μg | MT-9938 10μg | Placebo
Number analyzed (Participants) | 10 | 13 | 11 | 11
mm
  At 2 weeks | -8.77 (15.158) | -12.27 (12.154) | -6.56 (18.778) | -21.09 (26.719)
  At 4 weeks | -14.17 (22.631) | -19.46 (25.097) | -21.24 (20.300) | -23.63 (31.239)
  At 8 weeks (EOT) | -23.06 (23.686) | -29.16 (27.628) | -24.49 (42.732) | -30.09 (31.582)

3. Primary Outcome: Change From Baseline in Itch Severity Score
Description: The subject performed an assessment on day and nighttime symptoms of itch and effect of itch on sleep using a 5-point ordinal scale of itchiness (0 = none, 1 = mild, 2 = Moderate, 3=Severe, 4 = very severe). Assessments was made during each dialysis treatment (3x/week) and recorded on paper from the Screening Visit to the Follow-up Visit (Week 9). Change from Baseline (average over the Run-in Phase [Days -7 to -1]) in Weekly Averages of Itch Severity Score were assessed and score at 2, 4 and 8 weeks as specified in the protocol are reported. Amount of change score of plus indicates worsening, and minus indicates improvement.
Time Frame: 2 weeks, 4 weeks and 8 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MT-9938 2.5μg | MT-9938 5μg | MT-9938 10μg | Placebo
Number analyzed (Participants) | 10 | 13 | 11 | 11
score on a scale
  At 2 weeks | -0.77 (0.721) | -0.77 (0.542) | -0.43 (0.872) | -0.92 (1.106)
  At 4 weeks | -0.81 (0.835) | -1.08 (0.741) | -1.30 (0.885) | -0.90 (1.275)
  At 8 weeks (EOT) | -1.13 (1.003) | -1.49 (0.919) | -1.28 (1.094) | -1.28 (1.197)

4. Primary Outcome: Change From Baseline in Sleep Quality Assessment
Description: The PSQI has a minimum possible score of 0 (better sleep quality) and a maximum possible score of 10 (worse sleep quality). Subjects was asked to rate their sleep experience during the previous week. Pittsburgh Sleep Quality Index (PSQI) modified assessment was made during the dialysis treatment 1x/week every week and recorded on paper from the Screening Visit to the Follow-up Visit (Week 9).Change from Baseline (the Run-in Phase [Days -7 to -1]) were assessed and score at 2, 4 and 8 weeks as specified in the protocol are reported. Amount of change score of plus indicates worsening, and minus indicates improvement.
Time Frame: 2 weeks, 4 weeks and 8 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MT-9938 2.5μg | MT-9938 5μg | MT-9938 10μg | Placebo
Number analyzed (Participants) | 10 | 13 | 11 | 11
score on a scale
  At 2 weeks | -0.4 (1.06) | -0.2 (2.17) | -0.2 (1.64) | -1.0 (1.15)
  At 4 weeks | -0.4 (1.92) | -0.3 (1.65) | -1.1 (1.36) | -0.1 (1.36)
  At 8 weeks (EOT) | -1.1 (1.35) | -0.6 (1.62) | -1.2 (1.55) | -0.4 (1.59)

5. Primary Outcome: Change From Baseline in QoL Assessment (Skindex-10)
Description: The Skindex-10 has a minimum possible score of 0 (itching not bothersome) and a maximum possible score of 60 (itching very bothersome). The Skindex-10 is a self-administered questionnaire used to evaluate the health-related QoL in UP. It is comprised of 10 questions, adopted for pruritus from the Skindex-16, a widely used instrument for a variety of skin disease. Subjects was asked to identify on paper at Baseline and Weeks 2, 4, and 8 (EOT) what has bothered them most during the past week by marking along a scale 0 to 6 boxes from "never bothered" to "always bothered. Change from Baseline (the Run-in Phase [Days -7 to -1]) were assessed. Amount of change score of plus indicates worsening, and minus indicates improvement.
Time Frame: 2 weeks, 4 weeks and 8 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MT-9938 2.5μg | MT-9938 5μg | MT-9938 10μg | Placebo
Number analyzed (Participants) | 10 | 13 | 11 | 11
score on a scale
  At 2 weeks | -5.5 (8.55) | -11.6 (11.16) | -5.4 (9.27) | -13.6 (15.21)
  At 4 weeks | -0.5 (14.99) | -16.5 (15.00) | -16.4 (14.55) | -13.7 (17.68)
  At 8 weeks (EOT) | -11.9 (5.61) | -23.5 (15.52) | -19.2 (14.59) | -16.3 (14.63)

6. Primary Outcome: The Mean Value in Treatment Satisfaction (Patient's Global Impression of Change )
Description: The PGIC has a minimum possible score of 1 (very much improved) and a maximum possible score of 7 (very much worse). Subjects was asked to use a categorical scale with 7 categories to describe their global impression of change (PGIC) with study drug treatment. Subjects recorded their impression of change on paper at Weeks 2, 4, and 8 (EOT).
  Although the change from baseline (run-in phase [Days -7 to -1]) was specified as an outcome in this study, it was not calculated because the target enrollment was not met and no meaningful statistical analysis could be expected. Therefore, the mean value of patients at each point is shown instead.
Time Frame: 2 weeks, 4 weeks and 8 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MT-9938 2.5μg | MT-9938 5μg | MT-9938 10μg | Placebo
Number analyzed (Participants) | 10 | 13 | 11 | 11
units on a scale
  2 weeks | 3.1 (0.64) | 3.1 (1.51) | 3.0 (0.87) | 2.6 (1.07)
  4 weeks | 3.3 (0.71) | 2.8 (1.36) | 2.5 (0.93) | 2.8 (1.09)
  8 weeks | 2.6 (0.98) | 1.9 (0.90) | 2.1 (1.17) | 2.2 (1.30)

7. Primary Outcome: Change From Baseline in QoL Assessment (5-D-Itch Scale)
Description: The 5-D-Itch scale has a minimum possible score of 5 (better) and a maximum possible score of 25 (worse). Subjects was asked to assess QoL by means of the 5D-Itch-Scale at Baseline, Weeks 2, 4, and 8 (EOT). The 5D-Itch Scale is a 5-item (duration, degree, direction, disability, and distribution) multidimensional measure of pruritus itch. Change from Baseline (the Run-in Phase [Days -7 to -1]) were assessed. Amount of change score of plus indicates worsening, and minus indicates improvement.
Time Frame: 2 weeks, 4 weeks and 8 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MT-9938 2.5μg | MT-9938 5μg | MT-9938 10μg | Placebo
Number analyzed (Participants) | 10 | 13 | 11 | 11
score on a scale
  At 2 weeks | -2.8 (2.12) | -3.3 (2.46) | -3.0 (2.62) | -6.1 (5.84)
  At 4 weeks | -1.6 (4.17) | -5.1 (3.80) | -5.6 (3.16) | -5.7 (5.02)
  At 8 weeks | -3.7 (3.90) | -8.6 (4.25) | -6.2 (5.01) | -7.6 (4.53)

8. Primary Outcome: The Number of Patients in Excoriation
Description: Investigator and/or the designated medically qualified staff assessed the subject's excoriation at Baseline, and weekly thereafter, by completing the subject's answers to the following questions:
  Excoriation present? Yes/No If yes, please rate the severity: Mild/Moderate/Severe
  Although the change from baseline (run-in phase [Days -7 to -1]) was specified as an outcome in this study, it was not calculated because the target enrollment was not met and no meaningful statistical analysis could be expected. Therefore, the number of patients at each point is shown instead.
Time Frame: 2 weeks, 4 weeks and 8 weeks
Population: Not all rows could be analyzed with the overall number analyzed due to several reasons (e.g. patient discontinuation, missing data etc.), so some rows have different number of subjects analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | MT-9938 2.5μg | MT-9938 5μg | MT-9938 10μg | Placebo
Number analyzed (Participants) | 10 | 13 | 11 | 11
Participants
  Baseline: number analyzed (Participants) | 10 | 12 | 11 | 11
  Baseline: Excoriation not present | 7 | 6 | 7 | 7
  Baseline: Mild | 2 | 4 | 3 | 2
  Baseline: Moderate | 1 | 2 | 1 | 2
  Baseline: Severe | 0 | 0 | 0 | 0
  Baseline: Missing | 0 | 0 | 0 | 0
  2 weeks: number analyzed (Participants) | 8 | 12 | 9 | 10
  2 weeks: Excoriation not present | 6 | 7 | 7 | 7
  2 weeks: Mild | 2 | 5 | 2 | 3
  2 weeks: Moderate | 0 | 0 | 0 | 0
  2 weeks: Severe | 0 | 0 | 0 | 0
  2 weeks: Missing | 0 | 0 | 0 | 0
  4 weeks: number analyzed (Participants) | 8 | 13 | 8 | 10
  4 weeks: Excoriation not present | 6 | 11 | 7 | 7
  4 weeks: Mild | 2 | 2 | 1 | 2
  4 weeks: Moderate | 0 | 0 | 0 | 1
  4 weeks: Severe | 0 | 0 | 0 | 0
  4 weeks: Missing | 0 | 0 | 0 | 0
  8 weeks: number analyzed (Participants) | 7 | 12 | 9 | 9
  8 weeks: Excoriation not present | 6 | 9 | 9 | 7
  8 weeks: Mild | 1 | 2 | 0 | 1
  8 weeks: Moderate | 0 | 1 | 0 | 0
  8 weeks: Severe | 0 | 0 | 0 | 1
  8 weeks: Missing | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: The number of subjects with at least 1 treatment-emergent adverse event (TEAE). Please see the adverse event table for specific.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MT-9938 2.5μg | MT-9938 5μg | MT-9938 10μg | Placebo
Number analyzed (Participants) | 10 | 13 | 11 | 11
Participants | 6 | 5 | 9 | 6

ADVERSE EVENTS:
Time Frame: 8 weeks for treatment phase + 1 week follow-up visit after last dose
Arm/Group | MT-9938 2.5μg | MT-9938 5μg | MT-9938 10μg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/13 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 4/10 | 0/13 | 3/11 | 2/11
Other Adverse Events (participants affected / at risk) | 2/10 | 2/13 | 5/11 | 3/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-9938 2.5μg (N=10) | MT-9938 5μg (N=13) | MT-9938 10μg (N=11) | Placebo (N=11)
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pancreatitis Relapsing (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MT-9938 2.5μg (N=10) | MT-9938 5μg (N=13) | MT-9938 10μg (N=11) | Placebo (N=11)
Hyperprolactinaemia (Endocrine disorders) | 1 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 5 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PIs is that sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to sponsor for review. Sponsor can require changes to the communication which is considered confidential and/or proprietary. If necessary, sponsor shall have the right to request to delay the proposed disclosure for an additional 60 days.